CLINICAL TRIAL: NCT04450303
Title: Social Anxiety Telehealth Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tali Manber Ball, PhD, Instructor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56697
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Social Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Therapy (Experimental)
  Interventions: Behavioral: Telehealth CBT

INTERVENTIONS:
Behavioral: Telehealth CBT — The Coordinated Anxiety Learning and Management (CALM) program is an evidence-based, computer-assisted protocol for cognitive behavioral therapy (CBT) for anxiety, depression, and/or post-traumatic stress. CALM will be implemented via secure and HIPAA compliant video-conferencing software (enterprise Zoom), following modifications to address obstacles associated with physical distancing and the tele-health medium.
  Other Names: CALM

SUMMARY:
The COVID-19 pandemic has substantially increased the risk of adverse mental health outcomes; while physical distancing is required to reduce infection risk, it also increases loneliness and isolation and prevents access to traditional in-person therapy, which further contribute to risk of adverse mental health outcomes. These problems may be especially acute for individuals with social anxiety disorder (as many as 12% of Americans), however there is a limited evidence-base for telehealth options to directly address social anxiety. This project aims to adapt exposure therapy for social anxiety to a telehealth and physical distancing-compatible intervention, and test whether this effectively decreases loneliness in adults with elevated social anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+,
* Liebowitz Social Anxiety Scale (LSAS) total score > 50
* Fluent spoken and written English
* Access to the internet via a smartphone or computer with a camera
* Ability to provide informed consent.

Exclusion Criteria:

* History of mania or psychosis
* Moderate or severe substance use disorder within the past year
* Current psychiatric diagnosis of greater impairment than that arising from social anxiety
* High risk for suicide (>8 on the Mini International Neuropsychiatric Interview suicidality section)
* Prior exposure therapy (more than 2 sessions)
* Current psychotropic medication use
* Current psychotherapy other than couples counseling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | 12 weeks
  Social anxiety severity, lower scores are better (indicating less anxiety). Minimum score is 0, maximum score is 144.
Satisfaction with Therapy and Therapists Scale (STTS) | 12 weeks
  Therapy satisfaction subscale, higher scores are better (indicating greater satisfaction). Minimum score is 6, maximum score is 30.
UCLA Loneliness Scale version 3 | 12 weeks
  Loneliness, lower scores are better (indicating less loneliness). Minimum score is 20, maximum score is 80.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | 24 weeks
  Social anxiety severity, lower scores are better (indicating less anxiety). Minimum score is 0, maximum score is 144.
UCLA Loneliness Scale version 3 | 24 weeks
  Loneliness, lower scores are better (indicating less loneliness). Minimum score is 20, maximum score is 80.

CONTACTS AND LOCATIONS:
Overall Officials: Tali Ball, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided